CLINICAL TRIAL: NCT06332092
Title: A Phase 2, Randomized, Multicenter, Open-label, Study of FID-007 in Combination With Cetuximab in Patients With Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: FID-007 and Cetuximab in Treating Patients With Advanced Head and Neck Squamous Cell Carcinoma
Acronym: HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fulgent Pharma LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FID-007-003
Record Dates: First submitted 2024-03-12; First posted 2024-03-27 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: FID-007; Cetuximab; Paclitaxel; Head and Neck; p16
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Paclitaxel

STUDY DESIGN:
Intervention Model Description: Two different dosing regimens of FID-007 in combination with fixed-dose Cetuximab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Active Comparator): FID-007 (75 mg/m2) plus Cetuximab (500 mg/m2)
  Interventions: Drug: FID007
- Arm B (Active Comparator): FID-007 (125 mg/m2) plus Cetuximab (500 mg/m2)
  Interventions: Drug: FID007

INTERVENTIONS:
Drug: FID007 — Patients will receive FID007 via IV infusion at their assigned dose on Days 1, 8, and 15 of each 28-day cycle. Starting from Cycle 2, Cetuximab will be administered every 2 weeks on Days 1 and 15 of each 28-day cycle.
  Other Names: Paclitaxel in Polyethyloxazoline Polymer; FID-007; FID007 (CN); FID 007; Nanoencapsulated Paclitaxel FID-007

SUMMARY:
The goal of this FID-007 Clinical Trial is to compare the efficacy of different dosing regimens of FID-007 in combination with Cetuximab in patients with recurrent or metastatic Head and Neck Squamous Cell Carcinoma (HNSCC). The main questions it aims to answer are: to evaluate the efficacy, and to characterize the safety and tolerability. Eligible participants will be enrolled and randomized to 1 of 2 arms of FID-007 with fixed-dose Cetuximab in each 28-day cycle.

DETAILED DESCRIPTION:
The goal of this FID-007 Randomized, Multicenter, Open-label clinical trial is to compare the efficacy of different dosing regimens of FID-007 in combination with Cetuximab in patients with recurrent or metastatic Head and Neck Squamous Cell Carcinoma (HNSCC) based on objective response rate. The main questions it aims to answer are:

* To evaluate the efficacy of different dosing regimens of FID-007 in combination with Cetuximab in patients based on Best Overall Response (BOR), Duration of Response (DoR), Disease Control Rate (DCR), Progression-Free Survival (PFS), and Overall Survival (OS).
* To characterize the pharmacokinetics (PK) of FID-007 and its metabolites (6-α-hydroxypaclitaxel and 3'-p-hydroxypaclitaxel) following administration of different dosing regimens of FID-007 in combination with Cetuximab in patients with recurrent or metastatic HNSCC.
* To characterize the safety and tolerability of different dosing regimens of FID-007 in combination with Cetuximab in patients.

Eligible participants will be enrolled and randomized to 1 of 2 arms of FID-007 with fixed-dose Cetuximab (starting from Cycle 2, 500 mg/m2 intravenous [IV] infusion every 2 weeks on Days 1 and 15 of each 28-day cycle). Patients will receive FID-007 via IV infusion over 30 minutes at their assigned dose on Days 1, 8, and 15 of each 28-day cycle.

Patients will continue to receive Cetuximab and FID-007 until they meet the study drug discontinuation criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to provide informed consent before the start of any study-specific procedures.
2. Age ≥18 years old.
3. A diagnosis of recurrent or metastatic HNSCC at 1 of the following sites:

   1. Nasal/paranasal sinuses
   2. Nasopharynx (Epstein-Barr virus [EBV] negative only)
   3. Oral cavity
   4. Oropharynx
   5. Hypopharynx
   6. Larynx
4. Disease progression after treatment with PD-L1-based immune checkpoint inhibitor at any time. This can be as monotherapy or in combination with chemotherapy.
5. Measurable disease according to RECIST version 1.1.
6. Adequate treatment washout period of ≥21 days or 5 half-lives, whichever is shorter, for prior chemotherapy, radiotherapy, hormonal therapy, biological therapy, or immunotherapy before the first dose of study drug administration. Note: Palliative radiation is permitted but not ≤7 days before the first dose of study drug.
7. ECOG PS of 0 or 1.
8. Recovery from any toxic effects of previous chemotherapy, targeted therapy, or radiotherapy as judged by the investigator to Grade ≤1 (except for alopecia) according to NCI CTCAE version 5.0.
9. Adequate bone marrow and organ function defined as the following:

   Bone marrow function
   * Absolute neutrophil count ≥1500/mm3 (growth factor administration is not permitted ≤1 week before the screening assessment)
   * Platelet count ≥100,000/mm3 (platelet transfusion is not permitted ≤1 week before the screening assessment)
   * Hemoglobin ≥8 g/dL (criteria must be met without packed red blood cell transfusion ≤1 week before the screening assessment; chronic treatment with erythropoietin is permitted if the patient is on erythropoietin for ≥8 weeks)

   Blood clotting function

   • International normalized ratio (INR) ≤1.5 × upper limit of normal (ULN) and activated partial thromboplastin time ≤1.5 × ULN (except patients who are receiving therapeutic anticoagulation and whose INR should be within the therapeutic range)

   Renal function

   •Calculated clearance (using the Cockroft-Gault formula) ≥40 mL/min/1.73 m2. Actual body weight should be used for calculating creatinine clearance. For patients with a body mass index >30 kg/m2, lean body weight should be used instead

   Hepatic function
   * Total bilirubin ≤1.5 × ULN (patients with Gilbert's disease can have bilirubin >1.5 × ULN to <3 × ULN)
   * Aspartate aminotransferase/alanine aminotransferase ≤3 × ULN
10. An estimated life expectancy of at least 3 months based on investigator judgment.
11. Negative serum pregnancy test result at screening for female patients of childbearing potential.
12. Willingness to abide by the contraceptive requirements in Appendix 1 of the protocol.

Exclusion Criteria:

1. Known hypersensitivity to paclitaxel.
2. EBV-positive nasopharyngeal cancer, sinonasal undifferentiated carcinoma, esthesioneuroblastoma, or squamous cell carcinoma of the salivary gland or skin, based on the patient's medical history.
3. Received >1 prior line of anticancer therapy for recurrent or metastatic HNSCC. All patients must be previously treated with an immune checkpoint inhibitor either as monotherapy or in combination with chemotherapy. Patients treated with upfront combination chemo-immunotherapy followed by immunotherapy maintenance are considered to have received only 1 prior line of therapy. Chemotherapy given as part of treatment for locally advanced disease in the adjuvant or neoadjuvant setting is not considered a line of prior therapy for recurrent/metastatic disease. If the patient received prior treatment with Cetuximab, paclitaxel, or nab-paclitaxel in combination with radiation in the locally advanced setting and no relapse within 6 months of treatment discontinuation, enrollment is permitted if the treating physician believes that retreatment with Cetuximab or a taxane is a clinically reasonable option. However, patients who received these agents for recurrent or metastatic disease will be excluded.
4. Serious medical risk factors involving any of the major organ systems, or serious psychiatric disorders, that in the judgment of the investigator could compromise the patient's safety or the study data integrity.
5. Preexisting sensory neuropathy of Grade >1 severity by NCI CTCAE version 5.0 criteria.
6. Known history of uncontrolled HIV infection defined as CD4+ cells <350/mm3.
7. Requirement of systemic steroids at daily doses >10 mg prednisone equivalent systemic exposure daily, including for control of symptoms.
8. Use of any CYP2C8 and CYP3A4 inhibitor (eg, ketoconazole and other imidazole antifungals, erythromycin, fluoxetine, gemfibrozil, cimetidine, ritonavir, saquinavir, indinavir, and nelfinavir) or inducer (eg, rifampicin, carbamazepine, phenytoin, efavirenz, and nevirapine) in the previous 14 days before the first dose of study drug until the last PK sample is obtained in the study.
9. Known brain metastasis. Note: Patients whose central nervous system metastases have been treated by surgery or radiotherapy, who are no longer on corticosteroids, and who are neurologically stable are eligible.
10. Current or recent participation in a study of an investigational product in the prior 4 weeks. Note: Patients who have completed the treatment phase of an investigational study and have entered the follow-up phase of the investigational study may participate in FID-007-003 as long as it has been ≥4 weeks before the first dose of study drug.
11. Pregnancy, breastfeeding, or plans to become pregnant during the study or within 24 weeks after the last dose of study drug (Appendix 1 of the protocol).
12. Plans to donate/bank or retrieve eggs (ova, oocytes) during the study or within 24 weeks after the last dose of study drug (Appendix 1 of the protocol).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR assessed by Response Evaluation Criteria in Solid Tumors (RECIST) | Through study completion, an average of 1 year
  To evaluate the efficacy of different dosing regimens of FID-007 in combination with Cetuximab in patients with recurrent or metastatic HNSCC based on Objective Response Rate (ORR).

SECONDARY OUTCOMES:
BOR assessed by Response Evaluation Criteria in Solid Tumors (RECIST) | Through study completion, an average of 1 year
  Best Overall Response (BOR) measures the changes in tumor mass, growth (progression) or shrinkage (response) using the RECIST criteria.
Duration of Response (DoR) measurement | Through study completion, an average of 1 year
  The length of time that a tumor continues to respond to treatment without the cancer growing or spreading will be recorded.
Progression-free Survival (PFS) measurement | Through study completion, an average of 1 year
  The length of time to either radiological confirmed progression or death from any cause will be recorded.
Overall Survival (OS) measurement | Through study completion, an average of 1 year
  The length of time to death from any cause will be recorded.
Disease Control Rate (DCR) analysis | Through study completion, an average of 1 year
  The percentage of patients with advanced HNSCC who have achieved complete response, partial response and stable disease to different treatment regimens will be calculated.
Adverse Events (AEs) graded according to the CTCAE version 5.0 | Through study completion, an average of 1 year
  Safety and tolerability of different dosing regiments will be assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Vital Signs safety assessments | Through study completion, an average of 1 year
  Vital signs measurements include body temperature in Fahrenheit, respiratory rate, heart rate, and systolic and diastolic blood pressure measurements. Any confirmed, clinically significant abnormal vital sign measurements must be recorded as AEs.
Clinical Laboratory safety assessments | Through study completion, an average of 1 year
  Routine hematology, chemistry, and urinalysis to be performed at visits. Any confirmed, clinically significant abnormal laboratory results must be recorded as AEs.
ECGs safety assessment | Through study completion, an average of 1 year
  12-lead Electrocardiograms (ECGs) should be performed before the start and after the end of FID-007 infusion. An assessment of normal, clinically significant or abnormal, not clinically significant will be recorded.
Area Under the Plasma Concentration Versus Time Curve (AUC) of FID-007 | Cycle 2 (each cycle is 28 days)
  Application of pharmacokinetic principles to the safe and effective therapeutic management of drugs in an individual patient.
Peak Plasma Concentration (Cmax) | Cycle 2 (each cycle is 28 days)
  Application of pharmacokinetic parameters to the safe and effective therapeutic management of drugs in an individual patient.
Terminal/elimination half-life (t1/2) | Cycle 2 (each cycle is 28 days)
  Application of pharmacokinetic parameters to the safe and effective therapeutic management of drugs in an individual patient.
Clearance (CL) | Cycle 2 (each cycle is 28 days)
  Application of pharmacokinetic parameters to the safe and effective therapeutic management of drugs in an individual patient.
Volume of Distribution (Vd) | Cycle 2 (each cycle is 28 days)
  Application of pharmacokinetic parameters to the safe and effective therapeutic management of drugs in an individual patient.

CONTACTS AND LOCATIONS:
Overall Officials: Fulgent Clinical Sites, Principal Investigator — Fulgent Pharma LLC.
Locations (6):
- United States (6):
  - Highlands Oncology - North Hills, Fayetteville, Arkansas
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Moffitt Cancer Center Magnolia Campus, Tampa, Florida
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Northeast Texas Cancer & Research Institute, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lutz S. Ambulatory care keeps patients, hospitals on the move. Mod Healthc. 1989 Dec 1;19(48):20-2, 24, 28-32. No abstract available. PMID 10304137
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Burtness B, Rischin D, Greil R, Soulieres D, Tahara M, de Castro G Jr, Psyrri A, Brana I, Baste N, Neupane P, Bratland A, Fuereder T, Hughes BGM, Mesia R, Ngamphaiboon N, Rordorf T, Wan Ishak WZ, Ge J, Swaby RF, Gumuscu B, Harrington K. Pembrolizumab Alone or With Chemotherapy for Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma in KEYNOTE-048: Subgroup Analysis by Programmed Death Ligand-1 Combined Positive Score. J Clin Oncol. 2022 Jul 20;40(21):2321-2332. doi: 10.1200/JCO.21.02198. Epub 2022 Mar 25. PMID 35333599
- [Background] Burtness B, Goldwasser MA, Flood W, Mattar B, Forastiere AA; Eastern Cooperative Oncology Group. Phase III randomized trial of cisplatin plus placebo compared with cisplatin plus cetuximab in metastatic/recurrent head and neck cancer: an Eastern Cooperative Oncology Group study. J Clin Oncol. 2005 Dec 1;23(34):8646-54. doi: 10.1200/JCO.2005.02.4646. PMID 16314626
- [Background] Vermorken JB, Mesia R, Rivera F, Remenar E, Kawecki A, Rottey S, Erfan J, Zabolotnyy D, Kienzer HR, Cupissol D, Peyrade F, Benasso M, Vynnychenko I, De Raucourt D, Bokemeyer C, Schueler A, Amellal N, Hitt R. Platinum-based chemotherapy plus cetuximab in head and neck cancer. N Engl J Med. 2008 Sep 11;359(11):1116-27. doi: 10.1056/NEJMoa0802656. PMID 18784101
- [Background] Vermorken JB, Trigo J, Hitt R, Koralewski P, Diaz-Rubio E, Rolland F, Knecht R, Amellal N, Schueler A, Baselga J. Open-label, uncontrolled, multicenter phase II study to evaluate the efficacy and toxicity of cetuximab as a single agent in patients with recurrent and/or metastatic squamous cell carcinoma of the head and neck who failed to respond to platinum-based therapy. J Clin Oncol. 2007 Jun 1;25(16):2171-7. doi: 10.1200/JCO.2006.06.7447. PMID 17538161
- [Background] Fury MG, Sherman E, Lisa D, Agarwal N, Algazy K, Brockstein B, Langer C, Lim D, Mehra R, Rajan SK, Korte S, Lipson B, Yunus F, Tanvetyanon T, Smith-Marrone S, Ng K, Xiao H, Haque S, Pfister DG. A randomized phase II study of cetuximab every 2 weeks at either 500 or 750 mg/m2 for patients with recurrent or metastatic head and neck squamous cell cancer. J Natl Compr Canc Netw. 2012 Nov 1;10(11):1391-8. doi: 10.6004/jnccn.2012.0144. PMID 23138167
- [Background] Herbst RS, Kelly K, Chansky K, Mack PC, Franklin WA, Hirsch FR, Atkins JN, Dakhil SR, Albain KS, Kim ES, Redman M, Crowley JJ, Gandara DR. Phase II selection design trial of concurrent chemotherapy and cetuximab versus chemotherapy followed by cetuximab in advanced-stage non-small-cell lung cancer: Southwest Oncology Group study S0342. J Clin Oncol. 2010 Nov 1;28(31):4747-54. doi: 10.1200/JCO.2009.27.9356. Epub 2010 Oct 4. PMID 20921467
- [Background] Jain RK. Transport of molecules in the tumor interstitium: a review. Cancer Res. 1987 Jun 15;47(12):3039-51. PMID 3555767
- [Background] Baban DF, Seymour LW. Control of tumour vascular permeability. Adv Drug Deliv Rev. 1998 Oct 5;34(1):109-119. doi: 10.1016/s0169-409x(98)00003-9. PMID 10837673
- [Background] Serpe L. Conventional chemotherapeutic drug nanoparticles for cancer treatment. Kumar CS, ed. Nanomaterials for Cancer Therapy. Vol 6. Wiley-VCH Verlag GmbH & Co. KGaA, Weinheim; 2006:1-39.
- [Background] Desai N, Trieu V, Yao Z, Louie L, Ci S, Yang A, Tao C, De T, Beals B, Dykes D, Noker P, Yao R, Labao E, Hawkins M, Soon-Shiong P. Increased antitumor activity, intratumor paclitaxel concentrations, and endothelial cell transport of cremophor-free, albumin-bound paclitaxel, ABI-007, compared with cremophor-based paclitaxel. Clin Cancer Res. 2006 Feb 15;12(4):1317-24. doi: 10.1158/1078-0432.CCR-05-1634. PMID 16489089
- [Background] Grau JJ, Caballero M, Verger E, Monzo M, Blanch JL. Weekly paclitaxel for platin-resistant stage IV head and neck cancer patients. Acta Otolaryngol. 2009 Nov;129(11):1294-9. doi: 10.3109/00016480802590451. PMID 19863327
- [Background] Gibson MK, Li Y, Murphy B, Hussain MH, DeConti RC, Ensley J, Forastiere AA; Eastern Cooperative Oncology Group. Randomized phase III evaluation of cisplatin plus fluorouracil versus cisplatin plus paclitaxel in advanced head and neck cancer (E1395): an intergroup trial of the Eastern Cooperative Oncology Group. J Clin Oncol. 2005 May 20;23(15):3562-7. doi: 10.1200/JCO.2005.01.057. PMID 15908667
- [Background] Maghami E, Ismaila N, Alvarez A, Chernock R, Duvvuri U, Geiger J, Gross N, Haughey B, Paul D, Rodriguez C, Sher D, Stambuk HE, Waldron J, Witek M, Caudell J. Diagnosis and Management of Squamous Cell Carcinoma of Unknown Primary in the Head and Neck: ASCO Guideline. J Clin Oncol. 2020 Aug 1;38(22):2570-2596. doi: 10.1200/JCO.20.00275. Epub 2020 Apr 23. PMID 32324430
- [Background] Functional Assessment of Chronic Illness Therapy (FACIT) Group. Functional Assessment of Cancer Therapy - Head & Neck (FACT-HN), Version 4. Accessed September 12, 2023. https://www.facit.org/measures/FACT-HN
- [Background] [HMA] Heads of Medicines Agencies. Clinical Trial Facilitation Group page. Recommendations related to contraception and pregnancy testing in clinical trials. September 15, 2014. Accessed October 12, 2023. http://www.hma.eu/fileadmin/dateien/Human_Medicines/01-About_HMA/Working_Groups/CTFG/2014_09_HMA_CTFG_Contraception.pdf
- [Background] Yin R, Cheng T-C, Durst HD, Qin D. Enhancing Protein Activity through Nanoencapsulation. US Patent 6, 716, 450. 06-Apr-2004.
- [Background] Yin R, Durst HD, Emanuel PA, Hagnauer GL. Compositions and methods for enhancing bioassay performance through nanomanipulation. US Patent 6,773,928. August 10, 2004.
- [Background] Fulgent Pharma LLC. Investigator's Brochure for FID-007. Version 6. Fulgent Pharma, LLC; 2017.
- [Background] Erbitux- Cetuximab solution. Prescribing information. ImClone LLC; Revised: September 2021. https://uspl.lilly.com/erbitux/erbitux.html#pi